CLINICAL TRIAL: NCT04732247
Title: Evaluating Potential Benefits of Intranasal Oxytocin on Undersea Operator Training and Performance: Hyperoxic Swim-Induced Oxidative Stress and Inflammation
Brief Title: Oxytocin for Oxidative Stress and Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida Institute for Human and Machine Cognition (Other)
Collaborators: Office of Naval Research (ONR) (U.S. Federal Agency); University of Florida (Other); University of Alabama at Birmingham (Other); Translational Genomics Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-2020-0000
Record Dates: First submitted 2021-01-06; First posted 2021-02-01 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-06

CONDITIONS: Oxidative Stress; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized trial leveraging a wash-in design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All will remain blinded until completion of human subjects data collection except the research pharmacist providing intranasal oxytocin or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin nasal spray (Experimental): 4x per day (QID) intranasal treatment with oxytocin (48 IU per dose)
  Interventions: Drug: Oxytocin nasal spray
- Placebo nasal spray (Placebo Comparator): 4x per day (QID) intranasal treatment with placebo (identical to oxytocin nose spray minus the oxytocin)
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal treatment with oxytocin via nasal spray (48 IU per dose)
  Other Names: Oxytocin
  Arms: Oxytocin nasal spray
Drug: Placebo nasal spray — Intranasal treatment with placebo via nasal spray
  Other Names: Placebo
  Arms: Placebo nasal spray

SUMMARY:
Naval Special Warfare (NSW) operators are exposed to a variety of extreme environmental conditions and intense physical demands. In addition to breathing high pressure gases at depth, prolonged cold water immersion and inadequate recovery from sustained physical exertion negatively impact individual and team performance. Biotechnologies that could mitigate the effects of cold as well as support physical recovery represent a significant unmet need for the NSW operational community.

Oxytocin (OT) has a wide range of actions both locally in the brain and peripherally in the body including skeletal muscle. These peripheral effects can be mediated by classic ligand-receptor activation given the abundant expression of the oxytocin receptor in peripheral tissues, along with local expression of OT in peripheral tissues where it is likely to act in an autocrine manner. Exogenous OT via intranasal administration is FDA Investigational New Drug (IND)-approved and has been demonstrated as an easy and safe method to increase circulating OT concentrations that may augment actions on peripheral tissues.

Due to the pleiotropic effects of OT on whole body metabolism, thermogenesis, stress responses, pain, mood, inflammation, appetite, glycemic control, skeletal homeostasis, and skeletal muscle repair and regeneration, there is increasing interest in the administration of exogenous OT for benefits to human health, performance and resilience. However, the biological mechanisms by which OT exerts tissue-specific effects (e.g., skeletal muscle) remain poorly understood, particularly in humans. This project is designed to significantly advance this understanding while testing the central hypothesis that intranasally administered OT attenuates systemic and skeletal muscle oxidative stress and inflammation induced by the combined stressor of resistance swim exercise and hyperoxia.

DETAILED DESCRIPTION:
Naval Special Warfare (NSW) operators are exposed to a variety of extreme environmental conditions and intense physical demands. In addition to breathing high pressure and hyperoxic gases at depth, prolonged cold water immersion and inadequate recovery from sustained physical exertion negatively impact individual and team performance. Biotechnologies that could mitigate the effects of these extreme conditions as well as support physical recovery represent a significant unmet need for the NSW operational community.

Oxytocin (OT) has a wide range of actions both locally in the brain and peripherally including skeletal muscle and a number of peripheral targets. OT may attenuate acute cardiovascular stress responses, while chronic OT exposure may reduce risk of CVD and other chronic diseases via anti-inflammatory effects and attenuation of mitochondrial oxidative stress. These effects can be mediated by classic ligand-receptor activation given the abundant expression of the oxytocin receptor in peripheral tissues, along with local expression of OT in peripheral tissues where it is likely to act in an autocrine manner. Exogenous OT via intranasal administration is FDA Investigational New Drug (IND)-approved and has been demonstrated as an easy and safe method to increase circulating OT concentrations that may augment actions on peripheral tissues.

Due to the pleiotropic effects of OT on whole body metabolism, thermogenesis, stress responses, pain, mood, inflammation, appetite, glycemic control, skeletal homeostasis, and skeletal muscle repair and regeneration, there is increasing interest in the administration of exogenous OT for benefits to human health, performance and resilience. However, the biological mechanisms by which OT exerts tissue-specific effects (e.g., skeletal muscle) remain poorly understood, particularly in humans.

This project is designed to significantly advance this understanding while testing the central hypothesis that intranasally administered OT attenuates systemic and skeletal muscle oxidative stress and inflammation induced by the combined stressor of resistance swim exercise and hyperoxia. If efficacy is demonstrated, the ultimate deliverable would be an easily administered, adjunctive biological therapy expected to improve performance and resilience of undersea warfighters. The planned project will extend current IHMC research focused on developing biotechnologies to enhance human performance and resilience. The central hypothesis will be tested via two specific aims - using a rigorous, double-blind, placebo-controlled, randomized trial leveraging a wash-in design, enrolling N=40 18-39 y/o men.

Specific Aim 1. To investigate the efficacy of intranasal OT on attenuating systemic and skeletal muscle oxidative stress and inflammation induced by the combined stressor of intensive, resistance swim exercise and hyperoxia. Participants will be randomly assigned with a 1:1 distribution to 48 IU intranasal OT vs. placebo (saline). Investigators will test the effects of 4x per day (QID) intranasal treatment on performance and the acute inflammatory and oxidative stress responses to resistance swimming under hyperoxia, along with the timecourse of recovery over 48 h. To assess blood and muscle oxidative stress investigators will measure antioxidant enzymes, along with markers of oxidative stress-induced DNA damage, protein carbonylation, and lipid peroxidation. Systemic inflammation will be assessed via a 7-plex serum cytokine array, and muscle inflammation will be assessed via the TNF-a and IL-6 signaling pathways.

Specific Aim 2. To leverage proven molecular mapping strategies to identify key molecular transducers likely driving any effects of intranasal OT on systemic and muscle oxidative stress and inflammation throughout 48 h of recovery. Given the paucity of data on mechanisms by which exogenous OT exerts its effects, the investigators will take a discovery approach to identify novel molecular networks and pathways that are differentially regulated by OT vs. placebo during recovery from an intensive, resistance swim exercise under hyperoxia. To accomplish this the investigators will perform multi-level modeling that integrates data from metabolomics, transcriptomics (both long and small RNA sequencing from blood plasma and muscle), and miRNA sequencing of circulating extracellular vesicles (EVs).

If intranasal OT demonstrates efficacy, the deliverable would be an adjunctive biological therapy that mitigates oxidative stress as well as enhances performance during and recovery from resistance swimming under hyperoxia.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy (assessed via health, activity, and medical history)
* BMI < 30
* No chronic conditions that would preclude participation
* Recreationally skilled swimmer capable of a continuous 30 min kickboard swim

Exclusion Criteria:

- Regular smoking. The smoking exclusion includes all forms (cigarettes, vaping, etc) due to well-established effects on lung function and systemic oxidative stress and inflammation

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in muscle oxidative stress via glutathione reductase activity | Change in muscle glutathione reductase activity from before to 3 hours after the resistance swim + hyperoxia
  Change in muscle glutathione reductase enzyme activity assessed by measuring muscle tissue levels of the reduced product, glutathione (GSH)
Change in blood oxidative stress via glutathione reductase activity | Change in blood glutathione reductase activity from before to 3 hours after the resistance swim + hyperoxia
  Change in blood glutathione reductase enzyme activity assessed by measuring blood levels of the reduced product, glutathione (GSH)

SECONDARY OUTCOMES:
Change in systemic inflammation via serum concentration of interleukin-6 (IL-6) | Change in serum IL-6 concentration from before to 3 hours after the resistance swim + hyperoxia
  Change in systemic inflammation via serum concentration (pmol) of interleukin-6 (IL-6) assessed by enzyme-linked immunosorbent assay (ELISA)

OTHER OUTCOMES:
Change in muscle inflammation via muscle IL-6 pathway activity | Change in muscle STAT3 phosphorylation from before to 24 hours after the resistance swim + hyperoxia
  Change in muscle inflammation via muscle IL-6 pathway activity measured by phosphorylation state of STAT3 protein
Change in maximum aerobic power (VO2max) | Change in VO2max from before to 24 hours after the resistance swim + hyperoxia
  Change in VO2max (L/min) tested on a cycle ergometer using a maximal graded exercise protocol
Change in pulmonary function via spirometry | Before and 1 hour after the resistance swim + hyperoxia
  Change in pulmonary function via spirometry by measuring the maximum forced expiratory volume (L) expired in 1 second (FEV1)
Change in muscle soreness | Before and 24 hours after the resistance swim + hyperoxia
  Change in muscle soreness assessed using a visual-analog scale (VAS) with a continuous range from 0 (no soreness) to 10 (severe soreness)

CONTACTS AND LOCATIONS:
Overall Officials: Marcas M Bamman, PhD, Principal Investigator — Florida Institute for Human & Machine Cognition
Locations (3):
- United States (3):
  - Translational Genomics Research Institute, Phoenix, Arizona
  - University of Florida, Gainesville, Florida
  - Florida Institute for Human and Machine Cognition, Pensacola, Florida

IPD SHARING:
Plan to Share IPD: No
No IPD sharing planned